CLINICAL TRIAL: NCT02114736
Title: A Randomized Controlled Trial of Rectus Femoris Tenotomy Versus Botulinum Toxin A for Stiff Knee Gait After Stroke
Brief Title: Rectus Femoris Tenotomy Versus Botulinum Toxin A for Stiff Knee Gait After Stroke
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital of Mont-Godinne (Other)
Responsible Party: Principal Investigator, Deltombe Thierry, Professeur Clinique, University Hospital of Mont-Godinne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MG-SKG-57/2013
Record Dates: First submitted 2014-03-19; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Stroke; Spasticity
Keywords: Stroke; Muscle spasticity; Stiff knee gait; Botulinum toxin; Tenotomy
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Botulinum Toxins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rectus femoris tenotomy (Experimental): Surgical release of the proximal tendon of the rectus femoris
  Interventions: Procedure: Tenotomy of the proximal rectus femoris tendon
- Botulinum toxin in the rectus femoris muscle (Active Comparator): Botulinum toxin (200U Botox) injection in the rectus femoris muscle
  Interventions: Drug: Botulinum Toxin injection in the rectus femoris muscle

INTERVENTIONS:
Procedure: Tenotomy of the proximal rectus femoris tendon — Surgical release of the proximal tendon of the rectus femoris
  Other Names: Rectus femoris tenotomy
  Arms: Rectus femoris tenotomy
Drug: Botulinum Toxin injection in the rectus femoris muscle — Injections of 200U of Botox in the rectus femoris muscle with a 2ml/100U dilution
  Other Names: Rectus femoris botulinum toxin A injections
  Arms: Botulinum toxin in the rectus femoris muscle

SUMMARY:
Stiff knee gait is defined as the lack of knee flexion in the swing phase of gait. Stiff knee gait is a frequent condition among stroke patients leading to reduce gait speed and increase energy cost. In association with neuro-rehabilitation, botulinum toxin A injections in the rectus femoris is recommended. However, the botulinum toxin A effect is transient necessitating repeated injections.

The aim of this study is to compare the benefit of the rectus femoris tenotomy in comparison with botulinum toxin A injections according to the 3 domains of the International Classification of Functioning Disability and Health of the World Health Organisation

DETAILED DESCRIPTION:
INTRODUCTION

Stroke is the third cause of death and the leading cause of handicap among industrialized countries. Spasticity and co-contraction of the rectus femoris muscle following stroke is responsible for a lack of knee flexion in the swing phase of gait named stiff knee gait.

The rectus femoris spasticity is usually treated by oral medications, physical therapy and botulinum toxin A injections (1,2). As botulinum toxin A has a transient effect, injections must be repeated supporting to promote a permanent surgical treatment such as the rectus femoris tenotomy (3). However, no study has evaluate neither compare the effect of the rectus femoris tenotomy on gait and on the 3 domains of the International Classification of Functioning Disability and Health .

OBJECTIVE

To compare the effect of the rectus femoris tenotomy and of the botulinum toxin A injections for stiff knee gait after stroke according to the 3 domains of the International Classification of Functioning Disability and Health

METHODS

The investigators will recruited 20 chronic stroke patients presenting with stiff knee gait. The patients will be randomly assigned to a surgical group treated by rectus femoris tenotomy (10 patients) and to a medical group treated by rectus femoris botulinum toxin A injections.

Patients will be assessed before treatment, 2 months and 6 months after treatment by an assessor blinded therapist among the 3 domains of the International Classification of Functioning Disability and Health

PERSPECTIVE

The investigator hope to demonstrate the effectiveness of the rectus femoris tenotomy as a treatment of stiff knee gait after stroke

ELIGIBILITY:
Inclusion Criteria:

* stroke lasting for more than 6 months
* stiff knee gait
* rectus femoris spasticity (> Ashworth 2)
* transient improvement with previous botulinum toxine A injection in the rectus femoris
* stiff knee gait improved after rectus femoris diagnostic motor nere block
* able to walk on treadmill

Exclusion Criteria:

* pregnant women
* botulinum toxin A injections in the rectus femoris < 6 months
* previous surgery for stiff knee gait

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Ashworth scale at the rectus femoris | 6 months
  Spasticity assessment scale

SECONDARY OUTCOMES:
Stroke impairment assessment set (SIAS | 6 months
  Body function and structure scale for stroke patients
Tardieu scale | 6 months
  Spasiticty assessment scale
MRC (Medical research Council) scale | 6 months
  Muscle strength scale
Isometric muscle strenght assessment | 6 months
  Objective muscle strenght with isometric dynamometer
10 meter walking test | 6 months
  Gait speed assessment scale
Instrumented gait analysis | 6 months
  Kinetic and kinematic gait assessment in gait laboratory
ABILOCO scale | 6 months
  Activity level scale for gait validated according to Rasch model
EQ-5D-5L scale | 6 months
  Health quality of life scale

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Deltombe, M.D., Principal Investigator — University Hospital of Mont-Godinne, Université Catholique de Louvain
Locations (1):
- University Hospital of Mont-Godinne, Yvoir, Belgium

REFERENCES:
- [Background] Stoquart GG, Detrembleur C, Palumbo S, Deltombe T, Lejeune TM. Effect of botulinum toxin injection in the rectus femoris on stiff-knee gait in people with stroke: a prospective observational study. Arch Phys Med Rehabil. 2008 Jan;89(1):56-61. doi: 10.1016/j.apmr.2007.08.131. PMID 18164331
- [Background] Caty GD, Detrembleur C, Bleyenheuft C, Deltombe T, Lejeune TM. Effect of simultaneous botulinum toxin injections into several muscles on impairment, activity, participation, and quality of life among stroke patients presenting with a stiff knee gait. Stroke. 2008 Oct;39(10):2803-8. doi: 10.1161/STROKEAHA.108.516153. Epub 2008 Jul 17. PMID 18635841
- [Background] Namdari S, Pill SG, Makani A, Keenan MA. Rectus femoris to gracilis muscle transfer with fractional lengthening of the vastus muscles: a treatment for adults with stiff knee gait. Phys Ther. 2010 Feb;90(2):261-8. doi: 10.2522/ptj.20090151. Epub 2009 Dec 18. PMID 20023004